CLINICAL TRIAL: NCT00294502
Title: Antibiotic Lock Solutions in the Prevention of Catheter Related Bacteremia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3008
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2003-09

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Gentamicins; Citric Acid

INTERVENTIONS:
Drug: Gentamycin/citrate, Minocycline/EDTA

SUMMARY:
To study the efficacy of an antibacterial/anticoagulant solution instilled into the hemodialysis (HD) catheters after each treatment ("antibiotic lock solution - ALS") to prevent catheter related bacteremia (CRB) and to salvage catheters with established CRB.

DETAILED DESCRIPTION:
Scope of the problem. A large number of hemodialysis patients in this country rely on indwelling tunneled and non-tunneled catheters as vascular access for hemodialysis even though the K/DOQI guidelines discourage their use. In a study performed by ESRD network 11, [to which all Michigan dialysis centers submit data] 63% of patients initiated HD with a catheter as their sole form of vascular access. At 6 months after initiation of HD, 40% of these patients were still using a catheter. Other studies had shown that the prevalence of overall catheter use to be around 20% of all accesses.

Catheter associated infection. Current literature indicates that these catheters are associated with a disproportionate risk for infection, particularly CRB, resulting in high morbidity, mortality and healthcare expenditure. The 'epidemic' of ESRD in this country has seen an ever increasing reliance on these catheters not only to initiate the HD but also for long term treatment in those patients who have no other access options. It has been estimated that intravascular catheters are associated with more than 60,000 cases of nosocomial bacteremia each year. HD catheters pose a particularly high risk for developing infections because of their frequent use as well as their long-term use. All indwelling vascular catheters are colonized by micro-organisms within 24 hours after insertion. The deposition of biofilm on the external and internal surface of vascular catheters is thought to play an important role in the colonization process. The biofilm is produced by a combination of host factors (e.g., fibrinogen, fibrin, fibronectin and extracellular polysaccharides) and microbial products (e.g., glycocalyx or "slime").

Failure of antibiotics. Systemic antibiotics used to treat bacteremia do not penetrate catheter lumen and therefore do not eradicate the biofilm, leading to potential treatment failures and eventual sacrifice of the catheter. Recently published data suggests that using a combination solution with antibacterial/anticoagulant agents prevents the formation of the 'biofilm' in the catheter lumen thereby preventing CRB, as well as salvage the catheters in cases of established CRB. However, there continues to be a debate on the appropriate antibacterial agent as well as its optimal concentration, in order to eradicate a wide variety of organisms. Several other strategies were studied in the past 10 years to prevent CRB and CRI. These include eradication of nasal Staphylococcal carriage with mupirocin, using chlorhexidine for catheter hub cleaning and exit site disinfection and using mupirocin or Polysporin ointments to the exit site along with standard dressing. But emergence of antibiotic resistance as well as the high costs of administrating these methods continue to be barriers to their widespread use and cannot be relied upon to manage the high rate of infection by themselves.

Salvaging catheters. In the past, infected catheters were routinely removed, especially for Staphylococcus aureus infections, per the CDC guidelines. However, recent small studies indicate that strategies such as ALS packing or changing catheter over a guide wire can salvage a significant fraction of these catheters, thereby saving expense and morbidity, and preserving the site. Thrombotic occlusions and infection are the two most common complications of the HD catheters, each predisposing to the other. Some studies have shown that ALS packing has also improved the long-term catheter function by preventing the formation and propagation of the biofilm. Studying this aspect of catheter maintenance is also an important outcome for our proposed study.

Antibiotic Lock Solutions. We have identified 10 clinical trials (attached as appendix) in the published literature describing the results of antibiotic lock therapy for preventing infections in indwelling vascular catheters. All but one have demonstrated efficacy of ALS packing. Of the 9 successful trials, only 6 were randomized controlled trials and only 3 of these were done on HD catheters, as described below.

Need for a prospective study. If we can achieve the same superior results from our study incorporating the ALS packing strategy, we should be able to assess cost- effectiveness of using the ALS packing vs. standard approach as has been discussed in previous trials, but has not been systematically studied. In fact there are insufficient numbers of patients studies to even perform a meta-analysis. We feel that it is critical to prove the cost-effectiveness of the new strategy in order for it to be used in a widespread fashion.

The applicant, Anatole Besarab MD, has extensive experience in Nephrology and specifically in vascular access management. He has published, lectured, and coordinated symposia on vascular access care and is the current chair of the K/DOQI vascular access workgroup of the NKF.

This project is conceived for the following reasons.

* The CRB burden in the hemodialysis patients at this institution has reached overwhelming proportions and needs urgent strategies to counter this 'epidemic'. Current management guidelines rely mostly on treatment of established infections but do not aim at preventing these infections. This kind of economic burden and increased morbidity/mortality in patients are unacceptable in the current health care environment. Our study will add to the existing literature in defining the management guidelines for CRB.
* The Greenfield Health System (GHS) that provides dialysis care to the patients of the Henry Ford Health System includes several hundreds of patients and would be the ideal setting to study the proposed intervention. This population also represents a cross-section of many types of disease severity and number of co-morbid conditions. Therefore they provide an opportunity to observe the effects on the proposed intervention in different demographic settings.
* Henry Ford Hospital represents a completely new demography to study the effects of the proposed intervention. The disease burden with CRB in the population served by this area is higher than the national average and would be ideal to study the proposed intervention in more detail.
* The cost effectiveness of using the antibiotic lock therapy has not been well studied to date and will have a significant impact on the eventual formulation of treatment guidelines. In the setting of current economic burden in the health care industry, study of this issue is vital and timely. The vision of a simple, cheap intervention that can result in savings of millions of dollars is central to this study.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients with tunnelled catheters

Exclusion Criteria:

* patients on IV abx for infections, patients who have AV graft, AV fistulas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2004-05

PRIMARY OUTCOMES:
Incidence of symptomatic CRB

CONTACTS AND LOCATIONS:
Overall Officials: Antanole Bearabe, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Result] Allon M. Dialysis catheter-related bacteremia: treatment and prophylaxis. Am J Kidney Dis. 2004 Nov;44(5):779-91. PMID 15492943
- [Result] Dogra GK, Herson H, Hutchison B, Irish AB, Heath CH, Golledge C, Luxton G, Moody H. Prevention of tunneled hemodialysis catheter-related infections using catheter-restricted filling with gentamicin and citrate: a randomized controlled study. J Am Soc Nephrol. 2002 Aug;13(8):2133-9. doi: 10.1097/01.asn.0000022890.29656.22. PMID 12138146